CLINICAL TRIAL: NCT00190190
Title: Comparison of the Success Rate of a Procedure With Peeling of Limiting the Intern of the Retina Versus a Traditional Procedure Without Peeling of Limiting, at Patients Presenting a Macular Hole.
Brief Title: Internal Limiting Membrane Peeling for Large Macular Holes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Yannick VACHER, Department Clinical Research of Developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P040604; PS040604
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2008-07-18 (Estimated); Status verified 2007-07

CONDITIONS: Macular Hole
Keywords: Macular hole; internal limiting membrane; retina; surgery
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): With Peeling of Limiting the Intern of the Retina
  Interventions: Procedure: With Peeling of Limiting the Intern of the Retina
- 2 (Active Comparator): Traditional Procedure Without Peeling of Limiting
  Interventions: Procedure: Internal limiting membrane peeling

INTERVENTIONS:
Procedure: With Peeling of Limiting the Intern of the Retina — With Peeling of Limiting the Intern of the Retina
  Arms: 1
Procedure: Internal limiting membrane peeling — Traditional Procedure Without Peeling of Limiting
  Other Names: Traditional Procedure Without Peeling of Limiting
  Arms: 2

SUMMARY:
Rational of the study: for macular holes larger than 400 µm the rate of failure is of more than 20%. It is for these eyes that it is necessary to show the benefit of internal limiting membrane (ILM) peeling in term of vision and success rate. In order to test the benefit of this gesture, it is necessary to make a randomized study.

Primary objective: To show that the percentage of success (anatomical closing, confirmed by OCT) at third postoperative month is higher in the ILM peeling group.

Design of the study: Randomized multicentric study, in parallel groups, with individual benefit for the patient.

Tested Hypothesis: The success rate of the surgery of idiopathic macular holes larger than 400 µm is increased by the peeling of the MLI.

Awaited results: To show that the success rate of the surgery of idiopathic macular holes larger than 400 µm is improved by ILM peeling. This category could then have a success rate similar to the small holes. If this difference is not proven, it will remain no justification to continue this procedure which represents little risk but which is not either without consequence.

DETAILED DESCRIPTION:
Rational of the study: for macular holes larger than 400 µm the rate of failure is of more than 20%. It is for these eyes that it is necessary to show the benefit of internal limiting membrane (ILM) peeling in term of vision and success rate. In order to test the benefit of this gesture, it is necessary to make a randomized study.

Primary objective: To show that the percentage of success (anatomical closing, confirmed by OCT) at three postoperative months is higher in the ILM peeling group.

Design of the study: Randomized multicentric study, in parallel groups, with individual benefit for the patient.

Tested Hypothesis: The success rate of the surgery of idiopathic macular holes larger than 400 µm is increased by the peeling of the MLI.

Secondary objectives: - Percentage of success according to the effective success of peeling (failure, partial peeling, peeling 360°) in the peeling group of the MLI. - Gain of ETDRS visual acuity in the third postoperative month.- Progression of cataract - Frequency of the complications.

Number of subjects and duration of the study: 80 patients older than 18 yo , presenting a macular hole > 400 µm, divided into two parallel groups will be included and followed up 3 months. The estimated total duration of the study is 27 months.

Statistical analysis: The percentages of success in the 2 groups will be compared by a Chi ² or Fisher exact test. The test Q of COCHRAN will be used to take into account the ordered character of the categories.

Intermediate Analysis: An intermediate analysis is envisaged. The procedure of adjustment of the risk of Lan and DeMets will be used.

Awaited results: To show that the success rate of the surgery of idiopathic macular holes larger than 400 µm is improved by ILM peeling. This category could then have a success rate similar to the small holes. If this difference is not proven, it will remain no justification to continue this procedure which represents little risk but which is not either without consequence.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or higher than 18 years
* Patient presenting a TM idiopathic of stage 2, 3 or 4
* Macular hole > 400 µm in diameter
* Patient having been informed of the objectives and constraints of the study and having signed an informed consent

Exclusion Criteria:

* Patient age < 18 years.
* Patient having a strong myopia of the operated eye: correction carried or optimal >6 dioptres
* Patient MONOPHTHALMIA.
* Patient pseudophakia presenting an "insufficient" plan capsular CRYTALLINE.
* Patient presenting a cataract making impossible a good visualization of the bottom of eye.
* Patient presenting an important opacification capsular.
* Patient presenting an associated ocular pathology being able to interfere with the operation.
* Patient presenting a TM already operated of the eye to include

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
percentage of success (anatomical closing, confirmed by OCT) at third postoperative month, in both groups | at 3 months

SECONDARY OUTCOMES:
Percentage of success according to the effective success of peeling (failure, partial peeling, peeling 360°) in the peeling group of the MLI. | at 3 months
Gain of ETDRS visual acuity in the third postoperative month | at 3 months
Progression of cataract | at 3 months
Frequency of the complications. | at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ramin TADAYONI, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service d'Ophtalmolgie de l'Hôpital Lariboisière, Paris, France

REFERENCES:
- [Derived] Garcin T, Gaudric A, Sikorav A, Tadayoni R, Couturier A. Internal Limiting Membrane Peeling for Large Macular Holes Induces Only Structural Remodeling without Functional Impairment Over 12 Years. Ophthalmol Retina. 2025 Mar;9(3):253-262. doi: 10.1016/j.oret.2024.09.005. Epub 2024 Sep 12. PMID 39276867